CLINICAL TRIAL: NCT02413476
Title: Compared With Robotic-assisted and Laparoscopic-assisted Gastrectomy for Gastric Cancer on Surgical,Clinical and Oncological Outcomes
Brief Title: Comparison of Surgical,Clinical and Oncological Outcomes Between Robotic-assisted and Laparoscopic-assisted Gastrectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: wei bo (Other)
Responsible Party: Sponsor-Investigator, wei bo, Vice Director of the general surgery department, Chinese PLA General Hospital, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sample20152018
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-04

CONDITIONS: Gastric Cancer
Keywords: robotic-assisted gastrectomy; laparoscopic-assisted gastrectomy; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic-assisted Gastrectomy(RAG) (Experimental): Robotic-assisted Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Robotic-assisted Gastrectomy(RAG)
- Laparoscopic-assisted Gastrectomy(LAG) (Active Comparator): Laparoscopic-assisted Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic-assisted Gastrectomy(LAG)

INTERVENTIONS:
Procedure: Robotic-assisted Gastrectomy(RAG) — Surgical procedure will be performed with da vinci Surgical System.The type of reconstruction will be selected according to the surgeon's experience.
  Arms: Robotic-assisted Gastrectomy(RAG)
Procedure: Laparoscopic-assisted Gastrectomy(LAG) — Surgical procedure will be performed with laparoscopic techniques.The type of reconstruction will be selected according to the surgeon's experience.
  Arms: Laparoscopic-assisted Gastrectomy(LAG)

SUMMARY:
The study aims to compare the clinical outcomes between robotic-assisted and laparoscopic-assisted gastrectomy for gastric cancer,and evaluate the the feasibility and safety of robotic gastrectomy. Furthermore, the investigators can explore the patients who are more suitable for robotic gastrectomy.

DETAILED DESCRIPTION:
This is a prospective study lasting 36 months.

Minimally invasive gastrectomy is accepted widely in Asian countries. Laparoscopic-assisted gastrectomy offers improved early postoperative outcomes and improved long-term oncologic outcomes,but it still has its own limitations.The advantages of robotic surgery include a 3D imagine, convenient movements of the robotic arm, no tremor, and ambidextrous capability.

This study therefore aimed to compare the clinical results between robotic-assisted gastrectomy(RAG) using the da Vinci Surgical System and conventional laparoscopic-assisted gastrectomy(LAG) in gastric cancer patients.To evaluate the the feasibility and safety of robotic gastrectomy and explore the patients who are more suitable for robotic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven gastric cancer(early or advanced).
2. Age:older than 18 years old,younger than 80 years old.
3. cT1-4a(surgically resectable tumor),N0-3,M0 at preoperative evaluation according to the American Joint Committee on Cancer(AJCC) Cancer Staging Manual Seventh Edition
4. No obvious surgical contraindications.
5. American Society of Anesthesiology (ASA) score class I, II, or III
6. Written informed consent.

Exclusion Criteria:

1. Severe mental disorder
2. Pregnancy
3. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
4. History of previous gastrectomy,endoscopic mucosal resection or endoscopic submucosal dissection.
5. History of unstable angina or myocardial infarction within past six months
6. History of previous neoadjuvant chemotherapy or radiotherapy
7. History of other malignant disease within past 5 years.
8. Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
9. Any accompanying surgical condition needed to be performed in the same time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Five-year disease free survival rate | Up to 5 years post-operative

SECONDARY OUTCOMES:
Postoperative recovery course (time to first ambulation,flatus,liquid diet and soft diet,post-operative stay) | 7 days
  time to first ambulation,flatus,liquid diet and soft diet,post-operative stay
Complication (score based on the Clavien-Dindo classification system) | 30 days
  Compare the incidence,type and severity of early complications after gastrectomy,score based on the Clavien-Dindo classification system.
Mortality | 30 days
  Measured as 30-day mortality rate
Hospitalization expenses | 30 days
  the cost from admission to discharge
Quality of life | Up to 5 years post-operative
  The validated quality of life questionnaires EORTC QLQ-30 will be filled in pre-operative <5 days and post-operative at 6, 12, 24, 36, 48 and 60 months after surgery.
Five-year overall survival rate | Up to 5 years post-operative
Readmissions and recurrence rate | Up to 5 years post-operative
  The number of postoperative readmissions and recurrence rate.
Operating time | 1 day
  The operating time was defined as the time from skin incision to wound closure.
Intraoperative situation (The number of lymph node dissection,the number of positive lymph nodes,extra-cavity anastomosis time,intraoperative blood loss,the rate of conversion) | 1 day
  The number of lymph node dissection,the number of positive lymph nodes,extra-cavity anastomosis time,intraoperative blood loss,the rate of conversion

CONTACTS AND LOCATIONS:
Overall Officials: Wei bo, MD, Study Chair — Vice director of the general surgery department, Chinese PLA General Hospital

REFERENCES:
- [Background] Park JY, Ryu KW, Reim D, Eom BW, Yoon HM, Rho JY, Choi IJ, Kim YW. Robot-assisted gastrectomy for early gastric cancer: is it beneficial in viscerally obese patients compared to laparoscopic gastrectomy? World J Surg. 2015 Jul;39(7):1789-97. doi: 10.1007/s00268-015-2998-4. PMID 25670040
- [Background] Parisi A, Desiderio J. Establishing a multi-institutional registry to compare the outcomes of robotic, laparoscopic, and open surgery for gastric cancer. Surgery. 2015 Apr;157(4):830-1. doi: 10.1016/j.surg.2014.12.007. Epub 2015 Jan 26. No abstract available. PMID 25633739
- [Background] Lee J, Kim YM, Woo Y, Obama K, Noh SH, Hyung WJ. Robotic distal subtotal gastrectomy with D2 lymphadenectomy for gastric cancer patients with high body mass index: comparison with conventional laparoscopic distal subtotal gastrectomy with D2 lymphadenectomy. Surg Endosc. 2015 Nov;29(11):3251-60. doi: 10.1007/s00464-015-4069-1. Epub 2015 Jan 29. PMID 25631106
- [Background] Chuan L, Yan S, Pei-Wu Y. Meta-analysis of the short-term outcomes of robotic-assisted compared to laparoscopic gastrectomy. Minim Invasive Ther Allied Technol. 2015 Jun;24(3):127-34. doi: 10.3109/13645706.2014.985685. Epub 2014 Dec 3. PMID 25467019
- [Background] Suda K, Ishida Y, Uyama I. [Current status of robotic surgery for gastric cancer]. Gan To Kagaku Ryoho. 2014 Nov;41(11):1358-61. Japanese. PMID 25434438
- [Background] Huang KH, Lan YT, Fang WL, Chen JH, Lo SS, Li AF, Chiou SH, Wu CW, Shyr YM. Comparison of the operative outcomes and learning curves between laparoscopic and robotic gastrectomy for gastric cancer. PLoS One. 2014 Oct 31;9(10):e111499. doi: 10.1371/journal.pone.0111499. eCollection 2014. PMID 25360767
- [Background] Zong L, Seto Y, Aikou S, Takahashi T. Efficacy evaluation of subtotal and total gastrectomies in robotic surgery for gastric cancer compared with that in open and laparoscopic resections: a meta-analysis. PLoS One. 2014 Jul 28;9(7):e103312. doi: 10.1371/journal.pone.0103312. eCollection 2014. PMID 25068955
- [Background] Roviello F, Piagnerelli R, Ferrara F, Caputo E, Scheiterle M, Marrelli D. Assessing the feasibility of full robotic interaortocaval nodal dissection for locally advanced gastric cancer. Int J Med Robot. 2015 Jun;11(2):218-22. doi: 10.1002/rcs.1588. Epub 2014 Apr 15. PMID 24737464
- [Background] Son T, Lee JH, Kim YM, Kim HI, Noh SH, Hyung WJ. Robotic spleen-preserving total gastrectomy for gastric cancer: comparison with conventional laparoscopic procedure. Surg Endosc. 2014 Sep;28(9):2606-15. doi: 10.1007/s00464-014-3511-0. Epub 2014 Apr 3. PMID 24695982
- [Background] Junfeng Z, Yan S, Bo T, Yingxue H, Dongzhu Z, Yongliang Z, Feng Q, Peiwu Y. Robotic gastrectomy versus laparoscopic gastrectomy for gastric cancer: comparison of surgical performance and short-term outcomes. Surg Endosc. 2014 Jun;28(6):1779-87. doi: 10.1007/s00464-013-3385-6. Epub 2014 Jan 3. PMID 24385251
- [Background] Hyun MH, Lee CH, Kim HJ, Tong Y, Park SS. Systematic review and meta-analysis of robotic surgery compared with conventional laparoscopic and open resections for gastric carcinoma. Br J Surg. 2013 Nov;100(12):1566-78. doi: 10.1002/bjs.9242. PMID 24264778
- [Background] Marano A, Choi YY, Hyung WJ, Kim YM, Kim J, Noh SH. Robotic versus Laparoscopic versus Open Gastrectomy: A Meta-Analysis. J Gastric Cancer. 2013 Sep;13(3):136-48. doi: 10.5230/jgc.2013.13.3.136. Epub 2013 Sep 30. PMID 24156033
- [Background] Liao GX, Xie GZ, Li R, Zhao ZH, Sun QQ, Du SS, Ren C, Li GX, Deng HJ, Yuan YW. Meta-analysis of outcomes compared between robotic and laparoscopic gastrectomy for gastric cancer. Asian Pac J Cancer Prev. 2013;14(8):4871-5. doi: 10.7314/apjcp.2013.14.8.4871. PMID 24083761
- [Background] Kim HI, Park MS, Song KJ, Woo Y, Hyung WJ. Rapid and safe learning of robotic gastrectomy for gastric cancer: multidimensional analysis in a comparison with laparoscopic gastrectomy. Eur J Surg Oncol. 2014 Oct;40(10):1346-54. doi: 10.1016/j.ejso.2013.09.011. Epub 2013 Sep 17. PMID 24080199
- [Background] Hyun MH, Lee CH, Kwon YJ, Cho SI, Jang YJ, Kim DH, Kim JH, Park SH, Mok YJ, Park SS. Robot versus laparoscopic gastrectomy for cancer by an experienced surgeon: comparisons of surgery, complications, and surgical stress. Ann Surg Oncol. 2013 Apr;20(4):1258-65. doi: 10.1245/s10434-012-2679-6. Epub 2012 Oct 19. PMID 23080320
- [Background] Ortiz-Oshiro E, Exposito PB, Sierra JM, Gonzalez JD, Barbosa DS, Fernandez-Represa JA. Laparoscopic and robotic distal gastrectomy for gastrointestinal stromal tumour: case report. Int J Med Robot. 2012 Dec;8(4):491-5. doi: 10.1002/rcs.1456. Epub 2012 Aug 29. PMID 22930489